CLINICAL TRIAL: NCT06194526
Title: Whole Blood Transcriptomic Signal According to Coronary Atherosclerotic Plaque Burden Assessed by CT Angiography: CORPLAQ-TRAIT Pilot Study
Brief Title: Whole Blood Transcriptomic Signal According to Coronary Atherosclerotic Plaque Burden Assessed by CT Angiography
Acronym: CORPLAQ-TRAIT
Status: Enrolling by invitation | Type: Observational
Sponsor: MultiplAI Health Limited (Other)
Collaborators: Fundación para la Lucha contra las Enfermedades Neurológicas de la Infancia (Other)
Responsible Party: Sponsor
Other Study IDs: ACTC
Record Dates: First submitted 2023-10-31; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Calcific Coronary Arteriosclerosis; Coronary Stenosis; Coronary Plaque; Aortic Calcification; Atherosclerotic Plaque
Keywords: risk stratification; CVD screening; general population; transcriptomics; primary prevention; artificial intelligence; no history of CVD & history of CVD; subclinical; inflammation
MeSH Terms: conditions — Coronary Stenosis; Plaque, Atherosclerotic; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole-blood samples will be collected and analysed, and oral swab samples containing DNA will be stored for later analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present clinical study aims to identify transcriptomic patterns derived from whole blood samples related to coronary atherotic burden. Additionally, as a secondary analysis, the research team will explore the algorithm's ability to detect the presence of aortic disease and pro-inflammatory cardiometabolic alterations, such as hepatic steatosis and surrogate markers of coronary inflammation.

DETAILED DESCRIPTION:
This will be a prospective observational study. A convenience sample will be carried out to include 200 patients who attend the ENERI Medical Institute, La Sagrada Familia Clinic and Sanatorio Mendez with a clinical indication to be evaluated by a CCTA due to suspected CAD or known CAD. The study will have a baseline stage in which a clinical evaluation will be performed, blood samples will be drawn for transcriptome analysis and laboratory analysis. Then, a DNA sample obtained by swabbing the buccal mucose will be taken. Subsequently, the images obtained from the clinically indicated CCTA will be assessed to explore the outcomes of interest. At the end of patient enrollment, biological samples will be sequenced for in silico evaluation of the results. Finally, a 5-year follow-up will be carried out via telephone or email contact to collect data on the incidence of fatal and non-fatal cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 75 years, with a clinical indication to be evaluated by a CCTA due to suspected or known CAD.
* Signature of informed consent.

Exclusion Criteria:

* Previously known chronic renal or hepatic insufficiency.
* Active chronic lung disease, defined as: exacerbated asthma, exacerbated COPD, or pulmonary fibrosis.
* Myocardial infarction, unstable angina, cerebrovascular accident, or vascular interventions (any territory) in the past 6 months.
* Implantation of drug-eluting stents in the last 12 months.
* Revascularization surgery (By-pass)
* Indication of Angio-CT for congenital heart disease or Transcatheter Aortic Valve Replacement (TAVI)
* Presence/ diagnosis of heart failure symptoms or signs (ie. dyspnea, asthenia, edema) with objective evidence of pulmonary or systemic congestion at rest or with exercise in the last 6 months.
* Left ventricular ejection fraction <50% confirmed by objective diagnostic methods (eg doppler echocardiogram).
* Severe valvulopathies, confirmed by objective diagnostic methods (eg doppler echocardiogram).
* Uncontrolled hyper or hypothyroidism.
* Suprarenal insufficiency.
* Previous surgeries in the last 3 months.
* Severe trauma in the last 6 months, defined as one that involved bone fractures and/or surgical interventions.
* Known active cancer disease or under treatment (acute or preventive), or history of cancer disease without criteria for cure.
* Diagnosis of active autoimmune disease or any pathology under immunosuppressive treatment.
* Ongoing pregnancy, postpartum period of less than 12 months or breastfeeding.
* Other serious diseases with an estimated life expectancy of less than 12 months (according to the investigator's opinion).
* Temperature greater than 37.5°C recorded by a thermometer or any acute infection caused by viruses or bacteria confirmed by a health professional in the previous 30 days.
* Pacemaker/Cardio-Defibrillator Implantation.
* Prior to the study: heart rate > 70 l/m or atrial fibrillation or frequent extrasystoles that in the opinion of the specialist physician will affect the quality of the cardiovascular imaging.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200 Men and Women between 18 and 75 years of age with a physician's indication of a CCTA evaluation due to suspected or known CAD.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Coronary calcium score | At baseline (cross-sectional assessment)
  Coronary artery calcium (CAC) score (Agatston units) stratified with increasing risk according to the Society of Cardiovascular Computed Tomography Guidelines as CAC=0; CAC 1-99; CAC 100-299; and CAC≥300.
Total coronary plaque burden | At baseline (cross-sectional assesment)
  The extension of atherosclerotic disease burden will be assessed using the Modified Duke prognostic CAD index as follows: 1) ,50% stenosis; (2) ≥2 non-obstructive stenoses (including one artery with proximal disease or one artery with 50-69% stenosis); (3) two vessels with stenoses 50-69% or one vessel with ≥70% stenosis; (4) three-vessel disease with stenoses 50-69%, or two vessels ≥70%, or proximal LAD stenosis ≥70%; (5) three-vessel disease with stenoses ≥70% or two-vessel disease ≥70% with proximal LAD; (6) left main stenosis ≥50%.
Degree of coronary stenosis | At baseline (cross-sectional assesment)
  Each coronary segment will be graded based on the degree of coronary stenosis as 0% (no visible stenosis), 1-24% (minimal stenosis); 25-49% (mild stenosis); 50-69% (moderate stenosis); 70-99% (severe stenosis); 100% (occluded).
Coronary high-risk plaques (low-attenuation, positive remodeling; spotty calcification, or napkin-ring sign) | At baseline (cross-sectional assesment)
  Presence of any of the following features: low-attenuation (average density equal or lower than 30 Hounsfield units), positive remodeling (remodeling index equal or higher than 1.1; spotty calcification (average density >130 HU, diameter <3 mm in any direction with the length of the calcium <1.5 times the vessel diameter and width of the calcification less than two-thirds of the vessel diameter), or napkin-ring sign (ring-like attenuation pattern with peripheral high attenuation tissue that surrounds a central lower attenuation portion).

SECONDARY OUTCOMES:
Presence and extent of aortic calcification | At baseline (cross-sectional assessment)
  Aortic valve calcification score (Agatston units) as a continuous variable with increasing risk and without preestablished thresholds (ranging from 0 to 5.000 Agatston units).
Hepatic steatosis | At baseline (cross-sectional assessment)
  Defined as liver attenuation level lower than 48 Hounsfield units (HU), and lower than than the spleen attenuation.
Coronary artery inflammation (perivascular fat attenuation index) | At baseline (cross-sectional assessment)
  This secondary analysis will be performed using using specific software.
Death | Up to 5 years of Follow-up
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Rosana Poggio, MD MSc PhD, Principal Investigator — MultiplAI Health LTD
Locations (2):
- Argentina (2):
  - Sanatorio Julio Mendez, Ciudad Autónoma de Buenos Aire, Buenos Aires F.D.
  - Clinica Sagrada Familia, Ciudad Autónoma de Buenos Aire, Buenos Aires F.D.

DOCUMENTS (2):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT06194526/Prot_000.pdf
  • Informed Consent Form (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/26/NCT06194526/ICF_001.pdf